CLINICAL TRIAL: NCT07096310
Title: Comparison Between Carbapenems and Noncarbapenem Broad Spectrum Beta-lactam Antibiotics as Initial Antibiotic Therapy Against Sepsis in Burn Patients: A Prospective Study
Brief Title: Comparison Between Carbapenems and Noncarbapenem Beta-lactam Antibiotics in Septic Burn Patients
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ramy Mohamed Mohamed Abdelfattah, assistant lecturer of anesthesia and ICU, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD326/2023
Record Dates: First submitted 2025-07-04; First posted 2025-07-31 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Sepsis
Keywords: Meronem; Tazocin; sepsis; Burn
MeSH Terms: conditions — Sepsis; Burns | interventions — Meropenem; Piperacillin, Tazobactam Drug Combination; Piperacillin; Tazobactam

STUDY DESIGN:
Intervention Model Description: each drug will be given to every group according to dose according to Patient weight per KG
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Meronem group (Active Comparator): Meronem group will receive Meronem 2 gm Iv infusion over 3 hours every 8 hours per day
  Interventions: Drug: Meropenem I.V. 2g as a 3 hour infusion every 8 hours
- Tazocin group (Active Comparator): Tazocin group will receive non Carbapenems (Tazocin) 4.5 gm IV slow infusion over 20 minutes every 8 hours per day
  Interventions: Drug: Tazocin (pipercillin/tazobactam)

INTERVENTIONS:
Drug: Meropenem I.V. 2g as a 3 hour infusion every 8 hours — Non C group will receive non Carbapenems (Tazocin) 4.5 gm IV slow infusion over 20 minutes every 8 hours per day
  Other Names: Meronem
  Arms: Meronem group
Drug: Tazocin (pipercillin/tazobactam) — Non C group will receive non Carbapenems (Tazocin) 4.5 gm IV slow infusion over 20 minutes every 8 hours per day
  Other Names: Zocin
  Arms: Tazocin group

SUMMARY:
The aim of this work is to evaluate the efficacy associated with Meropenem(example of carbapenems) as initial therapy for sepsis in burn patients compared with Pipracillin/Tazobactam (example of non carbapenem beta lactam antibiotics).

DETAILED DESCRIPTION:
As causative pathogens are not usually identified at the time of initiating antibiotics in sepsis in burn patients, carbapenems are commonly used as an initial treatment. To reduce indiscriminate use of carbapenems, the efficacy of alternative empiric regimens, such as piperacillin-tazobactam and the fourth-generation cephalosporins, should be elucidated. The aim of this study is to compare efficacy of Meropenem and piperacillin tazobactam as an initial therapy of sepsis in burn patients .

ELIGIBILITY:
Inclusion Criteria:

* Burned patients admitted to Burn Unit of Ain Shams university hospitals diagnosed with sepsis, not transferred from other hospitals, Age group between 21 - 60 years old, ASA I and II.

Exclusion Criteria:

* Refusal of participation in the study,
* Patient with no signs of sepsis,
* Patients who died within 24 hours after admission,
* Patients concomitantly received carbapenems and other broad-spectrum beta-lactams,
* Data from the second and subsequent hospitalizations of patients who were hospitalized multiple times during the study period and used only the data from the first hospitalization,
* Patients younger than 21 years old and older than 60 years old.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to evaluate survival rate associated with carbapenems as initial therapy for sepsis in burn patients compared with non carbapenem antibiotics by comparing SOFA score between two groups. | 2 weeks
  The primary outcome of this work is to evaluate rate of survival associated with carbapenems as initial therapy for sepsis in burn patients compared with non carbapenem antibiotics by measuring SOFA score at day 4 and day 7 of starting of treatment.

SECONDARY OUTCOMES:
Occurrence rate of enterocolitis due to Clostridium difficile. (rate of patients with diarrhea and stool culture shows Clostridium difficile in each group). | 2 weeks
  Occurrence rate of enterocolitis due to Clostridium difficile.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Ali, MD, Study Chair — Ain Shams University; Osama R Abdelmalek, MD, Study Director — Ain Shams University; Thabet A Botros, MD, Study Director — Ain Shams University; Aya A Bayoumy, MD, Study Director — Ain Sham University
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Data Available with the corresponding author on visible request this is for patients privacy

REFERENCES:
- [Background] Rhodes NJ, Wagner JL, Davis SL, Bosso JA, Goff DA, Rybak MJ, Scheetz MH; MAD-ID Research Network. Trends in and Predictors of Carbapenem Consumption across North American Hospitals: Results from a Multicenter Survey by the MAD-ID Research Network. Antimicrob Agents Chemother. 2019 Jun 24;63(7):e00327-19. doi: 10.1128/AAC.00327-19. Print 2019 Jul. PMID 31061154
- [Background] Fleischmann-Struzek C, Mellhammar L, Rose N, Cassini A, Rudd KE, Schlattmann P, Allegranzi B, Reinhart K. Incidence and mortality of hospital- and ICU-treated sepsis: results from an updated and expanded systematic review and meta-analysis. Intensive Care Med. 2020 Aug;46(8):1552-1562. doi: 10.1007/s00134-020-06151-x. Epub 2020 Jun 22. PMID 32572531
- [Background] Ibrahim EH, Sherman G, Ward S, Fraser VJ, Kollef MH. The influence of inadequate antimicrobial treatment of bloodstream infections on patient outcomes in the ICU setting. Chest. 2000 Jul;118(1):146-55. doi: 10.1378/chest.118.1.146. PMID 10893372
- [Background] Umemura Y, Yamakawa K, Tanaka Y, Yoshimura J, Ogura H, Fujimi S. Efficacy of Carbapenems Compared With Noncarbapenem Broad-Spectrum Beta-Lactam Antibiotics as Initial Antibiotic Therapy Against Sepsis: A Nationwide Observational Study. Crit Care Med. 2023 Sep 1;51(9):1210-1221. doi: 10.1097/CCM.0000000000005932. Epub 2023 May 26. PMID 37232855
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Abe T, Ogura H, Shiraishi A, Kushimoto S, Saitoh D, Fujishima S, Mayumi T, Shiino Y, Nakada TA, Tarui T, Hifumi T, Otomo Y, Okamoto K, Umemura Y, Kotani J, Sakamoto Y, Sasaki J, Shiraishi SI, Takuma K, Tsuruta R, Hagiwara A, Yamakawa K, Masuno T, Takeyama N, Yamashita N, Ikeda H, Ueyama M, Fujimi S, Gando S; JAAM FORECAST group. Characteristics, management, and in-hospital mortality among patients with severe sepsis in intensive care units in Japan: the FORECAST study. Crit Care. 2018 Nov 22;22(1):322. doi: 10.1186/s13054-018-2186-7. PMID 30466493